CLINICAL TRIAL: NCT01149928
Title: Role of Cord Blood Hormones and Epinephrine in the Development of Transient Tachypnea of the Newborn
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Begum ATASAY, Ankara University School of Medicine, Department of Pediatrics
Other Study IDs: 08H3330006
Record Dates: First submitted 2010-06-21; First posted 2010-06-24 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2009-10

CONDITIONS: Wet Lung
Keywords: Fetal lung fluid; Pulmonary adaptation; Transient tachypnea of the newborn; Epinephrine; Stress hormones
MeSH Terms: conditions — Pulmonary Edema; Transient Tachypnea of the Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cord blood serum samples were stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- C/S delivered, wet lung
- C/S delivered, healthy infants

SUMMARY:
In this prospective, cross-sectional study, the aim was to investigate the possible role of cord stress hormones; adrenocorticotropic hormone (ACTH), cortisol, epinephrine, sT3, sT4, and thyroid-stimulating hormone (TSH) in the development of Transient Tachypnea of the Newborn (TTN), via their modulatory effect on epithelial sodium channels and Na-K-ATPase.

ELIGIBILITY:
Inclusion Criteria:

* Gestation age > 34 weeks
* C/S delivered infants
* Parental consent form signed

Exclusion Criteria:

* Gestation age < 34 weeks
* Maternal conditions that compromised fetal well-being (hypertensive disorder, diabetes, chorioamnionitis)
* Intrauterine growth retardation
* Congenital malformations
* Absence of parental consent

Ages: 34 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cesarean delivered, late preterm and term infants during the study period in Maternity Center of Ankara University
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Stress response at birth, as demonstrated by cord cortisol, adrenocorticotropic hormone, epinephrine, fT3, fT4, and thyroid-stimulating hormone in late preterm and term neonates developing transient tachypnea of the newborn. | postnatal first 24 hours
  At birth cord blood samples and perinatal data were collected from ceseraen deliveries of late preterm and term infants. Cord stress hormones of the infants with the diagnosis of TTN and gestational age matched controls were analyzed.

REFERENCES:
- [Derived] Atasay B, Ergun H, Okulu E, Mungan Akin I, Arsan S. The association between cord hormones and transient tachypnea of newborn in late preterm and term neonates who were delivered by cesarean section. J Matern Fetal Neonatal Med. 2013 Jun;26(9):877-80. doi: 10.3109/14767058.2013.765846. Epub 2013 Feb 8. PMID 23311764